CLINICAL TRIAL: NCT04827914
Title: Dissemination of an Inpatient Smoking Cessation Program to South Carolina Hospitals Study #1
Brief Title: Evaluation of an "Opt-Out" Inpatient Smoking Cessation Service on Smoking Behavior Study #1
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 107000
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enhanced Care Condition (Experimental)
  Interventions: Behavioral: Enhanced Care
- Basic Care Condition (Active Comparator)
  Interventions: Behavioral: Basic Care

INTERVENTIONS:
Behavioral: Enhanced Care — Smokers in the enhanced care group will receive live counseling (either in person or telehealth consult) while hospitalized combined with post-hospital discharge automated calls using interactive voice recognition (IVR) technology.
  Arms: Enhanced Care Condition
Behavioral: Basic Care — Smokers assigned to the basic care group will only receive the post-discharge IVR phone calls.
  Arms: Basic Care Condition

SUMMARY:
The modest goal of this study is to replicate the behavioral outcomes of the opt out MUSC-Tobacco Treatment Program in the following three patient groups: 1) psychiatric inpatients housed in the Institute of Psychiatry (IOP) in Charleston; 2) non-IOP patients seen in Charleston; and 3) patients seen in the other four MUSC affiliated hospitals combined (i.e., Chester, Florence, Lancaster, and Marion). The aims and the design/methods utilized for evaluation will be the same for each of the three patient groups.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years and older
* hospitalized cigarette smokers eligible for either enhanced or basic care
* discharged from the hospital back to their home

Exclusion Criteria:

* patients without a phone number
* those unable to communicate in the English language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1122 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Self-reported smoking prevalence 6-weeks after hospitalization. | Assessed 6-weeks post-discharge
  Hypothesize that patients exposed to the enhanced care intervention compared to basic care will report a 2-fold higher 7-day non-smoker prevalence rate after hospitalization (i.e., 20% vs 10%)
Self-reported use of FDA Approved Smoking Cessation Medication | Assessed 6-weeks post-discharge
  Hypothesize that patients exposed to the enhanced care intervention compared to basic care will report a 2.5-fold greater use of an FDA approved stop smoking medication after hospitalization (i.e., 20% vs 8%)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M Cummings, PhD, Principal Investigator — Medical University of South Carolina
Locations (6):
- United States (6):
  - Institute of Psychiatry, Charleston, South Carolina
  - MUSC, Charleston, South Carolina
  - MUSC, Chester, South Carolina
  - MUSC, Florence, South Carolina
  - MUSC, Lancaster, South Carolina
  - MUSC, Marion, South Carolina